CLINICAL TRIAL: NCT03396224
Title: Prospective Post Market Clinical Follow-up Study of the Avenir® Cemented Hip Stem
Brief Title: Avenir® Cemented Hip Stem - PMCF
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2013-03H
Record Dates: First submitted 2017-12-11; First posted 2018-01-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Primary Osteoarthritis; Post-Traumatic Osteoarthritis of Hip; Femoral Neck Fractures; Femoral Head Necrosis; Sequelae From Previous Hip Surgery; Osteotomies; Congenital Hip Dysplasia
Keywords: Total hip arthroplasty; Hip implant
MeSH Terms: conditions — Femoral Neck Fractures; Hip Dislocation, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Patients who received the Avenir® Cemented Hip Stem: Patients suffering from severe hip pain and disability requiring total hip arthroplasty and who meet the inclusion/exclusion criteria

SUMMARY:
The objective of this post-market clinical follow-up study is to confirm the safety and performance of the Avenir® Cemented Hip stem when used in primary total hip arthroplasty.

DETAILED DESCRIPTION:
This is a multicenter, prospective, non-controlled post-market clinical follow-up study to fulfill the post market surveillance obligations according to Medical Device Directive and MEDDEV 2.12-2.

The objectives of this study are to confirm the safety and performance of the Avenir Cemented Hip Stem when used in primary total hip arthroplasty at 6 weeks to 6 months, 1, 2, 3, 5, 7 and 10 years post-operatively.

The Avenir Cemented Hip Stem is a straight double-tapered stem offering 9 standard and 9 lateralized versions, the same as the uncemented version, the Avenir-Mueller Stem.

Safety will be evaluated by monitoring the frequency and incidence of adverse events and through radiographic review.

Performance will be based on the implant survival, overall pain and functional performances, subject quality-of-life and radiographic parameters of study subjects who received the Avenir® Cemented Hip stem.

Implant survival will be based on removal or intended removal of the device.

A total of 130 patients will be enrolled into the study at up to 4 sites.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age minimum.
* Patient is suffering from severe hip pain and disability requiring primary unilateral or bilateral total hip arthroplasty based on physical exam and medical history.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.

Exclusion Criteria:

* Patient is unwilling or unable to give consent, or to comply with the follow-up program.
* Acute, chronic, local, or systemic infections.
* Severe muscular, neural, or vascular diseases that endanger the limbs involved.
* Lack of bony structures proximal or distal to the joint, so that good anchorage of the implant is unlikely or impossible.
* Total or partial absence of the muscular or ligamentous apparatus.
* Any concomitant diseases that can jeopardize the functioning and the success of the implant.
* Allergy to the implanted material, especially to metal (e.g., stainless steel).
* Local bone tumors and/or cysts.
* Pregnancy
* Skeletal immaturity
* Patients who have any condition that would in the judgment of the Investigator place the patient at undue risk or interfere with the study. Any patient who is institutionalized, a known drug abuser or alcoholic or anyone who cannot understand what is required of them.
* Patients with plans to relocate during the study follow-up period.
* For patients biologically younger than 60 years with joint disease, a different reconstruction operation (e.g., osteotomy) or arthrodesis may be indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who:
  * are in need of a primary total hip arthroplasty
  * receive the Avenir® Cemented Hip Stem and compatible femoral head and acetabular cup
  * meet all the inclusion criteria and none of the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Implant survival based on removal or intended removal of the device and determined using the Kaplan-Meier method | 10 years

SECONDARY OUTCOMES:
The results of the hip surgery will be determined by the Harris Hip Score | 10 years
  The Harris Hip Score is a questionnaire filled by the surgeon with the patient who received a hip implant. The domains covered are pain, function, absence of deformity, and range of motion. The pain domain measures pain severity and its effect on activities and need for pain medication.
  The function domain consists of daily activities (stair use, using public transportation, sitting, and managing shoes and socks) and gait (limp, support needed, and walking distance). Deformity takes into account hip flexion, adduction, internal rotation, and extremity length discrepancy. Range of motion measures hip flexion, abduction, external and internal rotation, and adduction.
  There are 10 items. The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points).
The patient's quality-of-life will be determined by the EQ-5D score | 10 years
  EQ-5D is a standardized instrument for measuring health status. It is made up for two components.
  The description part: health status is measured in five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself. Usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have. In anxiety/depression dimension, it asks how anxious or depressed they are.
  Visual analogue scale: The patient marks his health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. The bottom rate (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine".
Abnormalities determined on X-rays in the bone region surrounding the implant will be reported | 10 years
Number of patient with adverse events related to the implant will be reported | 10 years
  Adverse events include: dislocations of the hip, revisions and removals of the implants

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (3):
- Cliniques Universitaires St-Luc UCL, Woluwe-Saint-Lambert, Brussels Capital, Belgium
- France (2):
  - Hôpital Gabriel Montpied - Service de chirurgie Orthopédique, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Hopital Lapeyronie - Service Orthopédie, Montpellier, Occitanie